CLINICAL TRIAL: NCT05457751
Title: The Effect of Orally Administered Metoprolol on the Frequency and Severity of Rocuronium Injection Pain
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozlem Sen, MD, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 20144
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- M: Group M: patients currently using metoprolol and who did not receive lidocaine before the application of rocuronium.
  Interventions: Procedure: Rocuronium injection pain
- ML: Group ML: patients currently using metoprolol and who received lidocaine before rocuronium application.
  Interventions: Procedure: Rocuronium injection pain
- L: Group L: patients currently not using metoprolol and received lidocaine before rocuronium application.
  Interventions: Procedure: Rocuronium injection pain
- C: Group C: patients currently not using metoprolol and who did not receive lidocaine before rocuronium application.
  Interventions: Procedure: Rocuronium injection pain

INTERVENTIONS:
Procedure: Rocuronium injection pain — 1: no reaction, 2: movement only in the ankle, 3: movement or withdrawal only in the arm (shoulder and ankle), 4: diffuse reaction (movement or withdrawal in more than one extremity, coughing and holding breath

SUMMARY:
In this study, we aimed to investigate the effect of metoprolol on the frequency and severity of pain caused by rocuronium injection in patients who started to use and were currently using oral metoprolol for any reason such as ischemic heart disease, hypertension, and arrhythmias. All patients were informed about the objectives of the study and gave informed written consent. The study was conducted in accordance with the relevant ethical principles of the Declaration of Helsinki. This study was planned as a prospective, placebo-controlled, cohort study were evaluated in four groups. Group M: patients currently using metoprolol and who did not receive lidocaine before the application of rocuronium. Group ML: patients currently using metoprolol and who received lidocaine before rocuronium application. Group L: patients currently not using metoprolol and received lidocaine before rocuronium application. Group C: patients currently not using metoprolol and who did not receive lidocaine before rocuronium application. 200 patients with 50 being in each of four groups were included in the study.

DETAILED DESCRIPTION:
Following the induction of general anesthesia with thiopental sodium, a researcher blind to the groups observed the pain during rocuronium injection based on the following scale:

1: no reaction, 2: movement only in the ankle, 3: movement or withdrawal only in the arm (shoulder and ankle), 4: diffuse reaction (movement or withdrawal in more than one extremity, coughing and holding breath).Heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), and SpO2 values were recorded before rocuronium administration, 1 and 3 minutes after rocuronium induction, and after intubation. Anesthesia maintenance was performed according to the discretion of the anesthetist. We checked the injection site regarding edema, rash, and thrombophlebitis after the first 24 hours of the operation.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years, ASA I-III, patients who received general anesthesia, patients who were using oral metoprolol for any reason such as ıschemic heart disease, arrhythmias.

Exclusion Criteria:

* Patients under 18 and above 75 years of age, with ASA IV class, those with known allergy to rocuronium and lidocaine, patients with chronic pain, pregnant women, those who had received analgesics or sedatives, and patients who were receiving calcium channel blocker that could affect pain were excluded from the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 200 patients, with 50 being in each group, were included in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2014-11-15 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Rocuronium injection pain | İntraoperative
  1: no reaction, 2: movement only in the ankle, 3: movement or withdrawal only in the arm (shoulder and ankle), 4: diffuse reaction (movement or withdrawal in more than one extremity, coughing and holding breath